CLINICAL TRIAL: NCT04590885
Title: Couple Communication Skills Training for Advanced Cancer
Brief Title: Coping Together: Couple-based Interventions for Cancer
Acronym: CCST2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00103232
Record Dates: First submitted 2020-10-09; First posted 2020-10-19 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-12

CONDITIONS: Advanced Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Couple Communication and Support (Other): CCST includes components to assist couples in communicating effectively, decreasing avoidance of important cancer-related issues, and providing each other with support. It includes training in skills for sharing one's thoughts and feelings and listening to one's partner and responding in a supportive manner, and joint problem solving. Participants will be asked to participate inactivities at home between sessions to strengthen skills acquisition.
  Interventions: Behavioral: Couple Communication Skills Training
- Healthy Lifestyle Informaion (Other): Healthy Lifestyle Information provides couples with health information relevant to cancer in a supportive environment. Sessions focus on the following topics: fatigue, sleep disturbance, nutrition, physical activity, survivorship care plans, and palliative care. Patients and partners are invited to discuss their experiences around the session topics with the therapist and ask questions about the information presented.
  Interventions: Behavioral: Healthy Lifestyle Information

INTERVENTIONS:
Behavioral: Couple Communication Skills Training — Participants attend six 60-minute sessions consisting of education and skills training to enhance cancer-related communication.
  Other Names: CCST
  Arms: Couple Communication and Support
Behavioral: Healthy Lifestyle Information — Participants attend attend six 60-minute sessions consisting of information and support across a range of cancer-related topics.
  Other Names: HLI
  Arms: Healthy Lifestyle Informaion

SUMMARY:
The objective of the proposed study is to evaluate the Couple Communication Skills Training (CCST) intervention in 250 patients with advanced cancer and their spouses/intimate partners. Couples will be randomized 1:1 to receive either the CCST or to an attention control condition (Healthy Living Information; HLI). We will evaluate CCST effects on a range of patient and partner relationship and psychological outcomes.

DETAILED DESCRIPTION:
For patients and their intimate partners, advanced cancer poses significant challenges that can negatively impact both individuals and the couple's collective well-being. Couples' ability to communicate openly and effectively with each other about cancer-related concerns can improve their psychological adjustment and quality of their relationship. Open and effective communication may also lead to better symptom management and goal-concordant care. However, many couples report difficulties communicating about cancer, even in the context of overall satisfying relationships. This can have a number of deleterious consequences, including deficits in emotional support, decreases in intimacy and relationship quality, and increased psychological distress. Thus, interventions designed to facilitate effective communication between cancer patients and their partners are likely to have beneficial effects on both individual and relationship functioning.

Prior research, including studies conducted by our team, has found that couple-based interventions that target communication lead to positive outcomes for cancer patients and their partners. However, most prior studies have been limited by reliance on an in-person treatment delivery format which keeps many couples from participating. In addition, prior studies have not targeted interventions to couples who are most likely to benefit. There is increasing evidence that psychosocial interventions for cancer, including couple-based interventions, should be targeted to those at risk of poor outcomes. Our prior research indicates that couples who report communication difficulties (e.g., high levels of holding back from discussing cancer-related concerns) have increased psychological distress and poorer relationship functioning and are most likely to benefit from a couple communication intervention specifically designed to addressed their communication problems.

The specific aims of this study are (1)To determine whether CCST significantly improves patients' and partners' individual psychological adjustment (i.e., psychological distress, life completion) and patient health and health care outcomes (physical well-being, symptom distress, advance care planning discussions and completion of advance directives, hospitalizations, and emergency department visits) compared to an education condition. (2) To determine whether, for couples receiving the CCST intervention, improvements in psychological adjustment, relationship functioning, and patient health are mediated by improvements in their communication, including objective measures of communication quality and communal coping (e.g., "we-talk") derived from couple conversations and self-reported protective buffering. (3) To examine differences in response to the CCST intervention for patients versus partners, for male versus female participants, and for patients with different cancer diagnoses (breast, lung, GI, GU). (4) To conduct an implementation-related process evaluation of the intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Married or in a committed intimate relationship
2. Diagnosis of one the following advanced cancers: Stage IIIB or IV non-small cell lung cancer or extensive stage small cell lung cancer, Stage III pancreatic cancer or Stage IV GI cancer, Stage IV GU cancer, Stage IV breast cancer and GYN cancer Stage III-IV ovarian, IV uterine, IV cervical.
3. Both members of the couple must speak and read English.
4. Patient and/or partner scores >=1.0 on the Holding Back screen.

Exclusion Criteria:

1. Patient lacks capacity for interview (documented diagnosis of active psychosis or dementia) or is unable to provide informed consent as assessed by research staff.
2. Patient has a life expectancy < 6 months as estimated by his/her treating oncologist.
3. Patient or partner is physically impaired in such a way that precludes the use of a computer or videoconferencing.
4. Patient or partner is too sick to participate, as judged by the oncologist or research staff.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440 (Actual)
Dates: Start 2020-10-20 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Changes in patient relationship functioning | Baseline, end of intervention (up to 8 months), 3 month post intervention follow-up
  Change in patient relationship satisfaction measured by the Couples Satisfaction Inventory (higher scores indicate higher satisfaction)
Changes in partner relationship functioning | Baseline, end of intervention (up to 8 months), 3 month post intervention follow-up
  Change in partner relationship satisfaction measured by the Couples Satisfaction Inventory (higher scores indicate higher satisfaction)
Changes in patient relationship functioning | Baseline, end of intervention (up to 8 months), 3 month post intervention follow-up
  Change in patient intimacy as measured by the Miller Social Intimacy Scale (higher scores indicate higher intimacy)
Changes in partner relationship functioning | Baseline, end of intervention (up to 8 months), 3 month post intervention follow-up
  Change in partner intimacy as measured by the Miller Social Intimacy Scale (higher scores indicate higher intimacy)

SECONDARY OUTCOMES:
Changes in patient psychological functioning | Baseline, end of intervention (up to 8 months), 3 month post intervention follow-up
  Change in patient psychological distress measured by the Hospital Anxiety and Depression Scale (higher scores indicate higher distress)
Changes in partner psychological functioning | Baseline, end of intervention (up to 8 months), 3 month post intervention follow-up
  Change in partner psychological distress measured by the Hospital Anxiety and Depression Scale (higher scores indicate higher distress)
Changes in patient psychological functioning | Baseline, end of intervention (up to 8 months), 3 month post intervention follow-up
  Change in patient mood as measured by the Positive and Negative Mood Scale (higher scores on the positive and negative mood subscales indicate higher negative and positive mood, respectively)
Changes in partner psychological functioning | Baseline, end of intervention (up to 8 months), 3 month post intervention follow-up
  Change in partner mood as measured by the Positive and Negative Mood Scale (higher scores on the positive and negative mood subscales indicate higher negative and positive mood, respectively)
Changes in patient psychological functioning | Baseline, end of intervention (up to 8 months), 3 month post intervention follow-up
  Change in patient life completion measured by the Life Completion scale of the QUAL-E (higher scores indicate higher completion)
Changes in partner psychological functioning | Baseline, end of intervention (up to 8 months), 3 month post intervention follow-up
  Change in partner life completion measured by the Life Completion scale of the QUAL-E Family (higher scores indicate higher completion)
Changes in patient psychological functioning | Baseline, end of intervention (up to 8 months), 3 month post intervention follow-up
  Change in patient physical well being as measured by the Physical Well Being subscale of the Functional Assessment of Cancer Therapy scale (higher scores indicate higher physical well being)
Changes in patient and partner psychological functioning | Baseline, end of intervention (up to 8 months), 3 month post intervention follow-up
  Change in symptom distress as measured by the Condensed Memorial Symptom Assessment Scale (higher scores indicate higher symptom distress)
Changes in patient psychological functioning | Baseline, end of intervention (up to 8 months), 3 month post intervention follow-up
  Change in patient advance care planning discussions (presence or absence, via patient self-report)
Changes in patient psychological functioning | Baseline, end of intervention (up to 8 months), 3 month post intervention follow-up
  Change in patient completion of advanced directives (presence or absence, via patient self-report)
Changes in patient psychological functioning | Baseline, end of intervention (up to 8 months), 3 month post intervention follow-up
  Change in patient hospitalizations (number of hospitalizations per patient self-report, validated by medical record review)
Changes in patient psychological functioning | Baseline, end of intervention (up to 8 months), 3 month post intervention follow-up
  Change in patient emergency department visits (number of emergency department visits per patient self-report, validated by medical record review)

CONTACTS AND LOCATIONS:
Overall Officials: Laura Porter, PhD, Principal Investigator — Duke
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Porter LS, Ramos K, Baucom DH, Steinhauser K, Erkanli A, Strauman TJ, Zafar SY, Check DK, Leo K, Liu E, Keefe FJ. Evaluating a couple communication skills training (CCST) intervention for advanced cancer: study protocol for a randomized controlled trial. Trials. 2022 Aug 26;23(1):712. doi: 10.1186/s13063-022-06656-4. PMID 36028908

DOCUMENTS (1):
  • Informed Consent Form (2023-10-30): https://cdn.clinicaltrials.gov/large-docs/85/NCT04590885/ICF_000.pdf